CLINICAL TRIAL: NCT03471780
Title: The Importance of Transperineal US in Labour
Brief Title: Evaluation of Transperineal US in Labour
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Assistant Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: labour US
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Labor Long
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound — Transperineal us are made to pregnant ladies in labour

SUMMARY:
Assessment of progress of labour is an important step in decision making of obstetricians

DETAILED DESCRIPTION:
delayed progress of labour resemble an annoying problem to obstetrician so noninvasive diagnostic methods can play an important role in implementing a guidelines to follow patients in labour as transperineal US .

ELIGIBILITY:
Inclusion Criteria:

* pregnant women in labour
* Full term

Exclusion Criteria:

* pregnant ladies not in labour
* Preterm labour

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women in labour
Study Population: * pregnant women in labour
  * Full term
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-04-10 (Estimated); Study Completion 2019-04-10 (Estimated)

PRIMARY OUTCOMES:
the number of participants who will deliver by normal delivery | within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
no plan is decided now